CLINICAL TRIAL: NCT06402669
Title: Time to Hospitalization and Limb Loss in Blunt Extremity Trauma
Brief Title: Extremity Trauma At a Level 1 Trauma Center
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-04
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-05

CONDITIONS: Trauma Injury; Trauma Blunt; Vascular Trauma
MeSH Terms: conditions — Accidental Injuries; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Transferred from Outside Hospital: Patients with blunt or penetrating trauma that are transferred from an outside hospital to admitting level 1 trauma center
  Interventions: Other: Packed Red Blood Cell Administration
- Direct Admission to Hospital: Patients with blunt or penetrating trauma that are directly brought to level 1 trauma center
  Interventions: Other: Packed Red Blood Cell Administration

INTERVENTIONS:
Other: Packed Red Blood Cell Administration — Difference in occurrence of mortality in patients transferred versus directly admitted who have packed red blood cell administration in the first four hours of arrival to the hospital.

SUMMARY:
Blunt vascular trauma to the lower extremity has been associated with injuries to the anteroposterior tibial arteries or popliteal artery in the form of transection, occlusion, or intimal injury. With many blunt injuries resulting in orthopedic fractures, the incidence of limb loss increases substantial. Distal vascular injuries combined with complex orthopedic fractures are more likely to result in limb loss. A recent retrospective study showed two main predicative factors resulting in limb loss was a result of multi-segmental bone fractures and prolong ischemic time greater then 10 hours.

DETAILED DESCRIPTION:
Extremity trauma continues to remain a notable cause for presentation to the emergency department for trauma-level care, with penetrating extremity injuries comprising 5 to 15% of trauma cases. In the setting of vascular extremity injury, appropriate care protocols must be established to prevent life threatening complications including infection, non-union, limb salvage failure, and death. The two primary mechanisms of extremity trauma include penetrating trauma involving projectile and stab injuries, as well as blunt trauma involving fractures and joint dislocations. While central or peripheral vascular injuries constitute 1-2% of traumatic injuries, they result in more than 20% of trauma-related mortality demonstrating the importance of timely and efficacious care of extremity trauma patients, with particular emphasis on vascular injury assessment. The health care facility settings in which patients present have significant implications in the level of care provided, as availability of diagnostic and therapeutic resources may be limited in some settings. In such circumstances, patients may be transferred to alternate care facilities for higher level of care, with timing of transfer playing a substantial role in successful trauma patient care.

While it is noted that the treatment of severely injured patients in higher level trauma centers allows for access to increased care resources and improved prognostic outcomes, the patient outcomes of trauma patients transferred from lower level to higher level trauma centers may not be as clear. With regards to interhospital patient transfers, there are established statewide trauma policies that guide "re-triage," which is defined as the urgent or emergent transfer of critically ill trauma patients from a non-trauma or lower level trauma facility to an upper level trauma center for higher level of care. The categories for re-triage consideration include perfusion, respiratory status, neurologic status, anatomic findings, and provider judgment. For example, anatomic findings that necessitate transfer to higher level of care facilities include extremity injury with neurovascular compromise. Important components of re-triage include early identification of patients who require higher levels of care as well as established transfer agreements between sending and receiving care facilities. Recognizing that patient transfers may impact overall health outcomes such that transferred extremity trauma patients may have worse clinical outcomes compared to non-transferred patients, the investigators aim to investigate the relationship between transfer status and patient outcomes through conducting a retrospective observational case-control review of extremity trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or higher with blunt or penetrating extremity trauma injuries

Exclusion Criteria:

* Pregnant females with blunt or penetrating extremity trauma injuries
* Catastrophic head injuries
* Individuals discharged from the hospital in the first 24 hours of being seen

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was completed at the Arrowhead Regional Medical Center (ARMC) in San Bernardino County, California. The ARMC is a 456-bed acute-care teaching facility and ACS-verified level I trauma center. The ARMC emergency department (ED) is one of the busiest in the state of California with more than 100,000 visits and over 3,000 adult trauma cases annually.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Measured in the first 30 days of admission
  Incidence of mortality associated with transfer status
Length of total hospital stay | Length of total hospital stay from admission in the hospital is defined as the time frame between admission and discharge. The time frame of collection until the event occurred was 180 days.
  The time spent hospitalized in days.
Operative Cases | Time frame is from admission to discharge and would be collected in the first 180 days.
  The total operative cases required for a patient
Admission lactate levels | he estimated period of time over which preoperative lactate levels are measured occur in the initial 2 hours after admission to the hospital
  Admission lactate levels were defined as the first measured lactate level on admission of an individual who presented as a trauma patient.

CONTACTS AND LOCATIONS:
Overall Officials: Aldin Malkoc, Study Chair — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devendra A, Nishith P G, Dilip Chand Raja S, Dheenadhayalan J, Rajasekaran S. Current updates in management of extremity injuries in polytrauma. J Clin Orthop Trauma. 2021 Jan;12(1):113-122. doi: 10.1016/j.jcot.2020.09.031. Epub 2020 Sep 24. PMID 33716436
- [Background] Waalwijk JF, Lokerman RD, van der Sluijs R, Fiddelers AAA, den Hartog D, Leenen LPH, Poeze M, van Heijl M; Pre-hospital Trauma Triage Research Collaborative (PTTRC). The influence of inter-hospital transfers on mortality in severely injured patients. Eur J Trauma Emerg Surg. 2023 Feb;49(1):441-449. doi: 10.1007/s00068-022-02087-7. Epub 2022 Sep 1. PMID 36048180
- [Background] Garwe T, Cowan LD, Neas B, Cathey T, Danford BC, Greenawalt P. Survival benefit of transfer to tertiary trauma centers for major trauma patients initially presenting to nontertiary trauma centers. Acad Emerg Med. 2010 Nov;17(11):1223-32. doi: 10.1111/j.1553-2712.2010.00918.x. PMID 21175521
- [Background] Staudenmayer KL, Hsia RY, Mann NC, Spain DA, Newgard CD. Triage of elderly trauma patients: a population-based perspective. J Am Coll Surg. 2013 Oct;217(4):569-76. doi: 10.1016/j.jamcollsurg.2013.06.017. PMID 24054408